CLINICAL TRIAL: NCT02154178
Title: Fungal Biomarkers to Reduce Duration of Empirical Antifungal Therapy: a Randomized Comparative Study
Brief Title: Fungal Biomarkers to Reduce Duration of Empirical Antifungal Therapy: a Randomized Comparative Study (STAFE)
Acronym: STAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012_53; 2013 A00756 39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2014-05-24; First posted 2014-06-03 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2017-03

CONDITIONS: Fungal Infection; Critical Illness
Keywords: empiric antifungal therapy; biomarkers; invasive fungal infection; Candida
MeSH Terms: conditions — Mycoses; Critical Illness; Invasive Fungal Infections; Torulopsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biomarker group (Experimental): Intervention group, in which the duration of empirical antifungal therapy will be based on the results of biomarkers.
  Biomarker group
  Interventions: Other: Biomarker group
- Control group (No Intervention): Control group, in which the duration of empirical antifungal therapy will be based on international recommendations (14 days).

INTERVENTIONS:
Other: Biomarker group — use of invasive fungal disease biomarkers (β-1,3-glucan, mannan/anti-mannan antibodies)
  Other Names: intervention group
  Arms: Biomarker group

SUMMARY:
The investigators hypothesized that the use of biomarkers of invasive fungal infections would increase the percentage of early discontinuation of empirical antifungal therapy and thus reduce the duration of treatment in ICU patients.

DETAILED DESCRIPTION:
The duration of empirical/preemptive anti fungal treatment will be based in the intervention group on biomarker results.

Biomarkers of fungal disease will performed before starting anti fungal treatment and at day 4.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Patients requiring empiric antifungal therapy the first time in the ICU
* Predictable duration of hospitalization in the ICU ≥ 6 days

Exclusion Criteria:

* Neutropenia (WBC <1000 or neutrophils <500/mm3)
* Immunosuppressive therapy (chemotherapy within 3 months prior to the ICU admission, solid organ graft under immunosuppressive therapy)
* invasive fungal infection documented in the three previous months
* Antifungal treatment in the three previous months
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
percentage of early discontinuation of empiric antifungal therapy | 7 days
  Early discontinuation is defined as discontinuation of anti fungal treatment before the 7th day after the start of treatment

SECONDARY OUTCOMES:
mortality in ICU | 28 days after ICU admission
  death during the 28 days following ICU admission
duration of mechanical ventilation and ICU stay | 28 days after ICU admission
  mechanical ventilation duration during the 28 days following ICU admission
fungal colonization / infection after antifungal therapy, with or without resistant strains | 28 days after ICU admission
  Any fungal colonization or infection diagnosed during the 28 days following ICU admission
the cost of the antifungal therapy on a per duration prescribe | 28 days after ICU admission
the cost of hospital stays | 28 days after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD, PhD, Principal Investigator — Univ Hosp of Lille, France
Locations (1):
- ICU, Salengro Hospital, University Hospital of Lille, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rouze A, Loridant S, Poissy J, Dervaux B, Sendid B, Cornu M, Nseir S; S-TAFE study group. Biomarker-based strategy for early discontinuation of empirical antifungal treatment in critically ill patients: a randomized controlled trial. Intensive Care Med. 2017 Nov;43(11):1668-1677. doi: 10.1007/s00134-017-4932-8. Epub 2017 Sep 22. PMID 28936678